CLINICAL TRIAL: NCT02108327
Title: Comparison of Blood Loss Between Surgical Blade and Unipolar Electrocautery in Primary Total Knee Arthroplasty
Brief Title: Blood Loss Between Surgical Blade and Unipolar Electrocautery in TKA
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, principal investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: orthoTU07
Record Dates: First submitted 2014-04-01; First posted 2014-04-09 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Blood Loss
Keywords: Blood loss; total knee arthroplasty; hot knife; cold knife; unipolar electrocautery; surgical blade
MeSH Terms: conditions — Hemorrhage | interventions — Electrocoagulation; Conization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgical blade (Experimental)
  Interventions: Procedure: surgical blade
- Unipolar electrocautery (Active Comparator)
  Interventions: Procedure: electrocautery

INTERVENTIONS:
Procedure: surgical blade — Using surgical blade all the time of surgery
  Other Names: hot knife
  Arms: surgical blade
Procedure: electrocautery — Using electrocautery all the time except at skin incision
  Other Names: cold knife
  Arms: Unipolar electrocautery

SUMMARY:
Using of surgical blade may have less blood loss than unipolar electrocautery in Total Knee Arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee who undergoing unilateral primary total knee arthroplasty
* age 50-85 years old
* ASA class 1-3

Exclusion Criteria:

* unable to perform spinal anaesthesia
* history of coagulation disorder
* renal impairment (CrCl <30 mL/min) or cirrhosis
* platelet count < 100,000 or abnormal coagulogram
* on pacemaker
* stop anti-platelet or anti-coagulogram less than 7 days

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Blood loss | 48 hours
  - detected total blood loss from hemoglobin at 24,48 hours after surgery, maximum Hb drop and blood loss collected in radivac drain

SECONDARY OUTCOMES:
inflammation | 48 hours
  determine inflammatory response with C-rective protein (CRP) at post-op 48 hours
Knee function | 3 months
  measured with WOMAC
knee range of motion | 3 months
complication | 2 weeks
  detected with wound dehiscence, wound infection

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic department, Faculty of medicine, Thammasat university, Klongluang, Changwat Pathum Thani, Thailand

REFERENCES:
- [Derived] Tammachote N, Kanitnate S. Electric cautery does not reduce blood loss in primary total knee arthroplasty compared with scalpel only surgery a double-blinded randomized controlled trial. Int Orthop. 2018 Dec;42(12):2755-2760. doi: 10.1007/s00264-018-4048-y. Epub 2018 Jul 3. PMID 29968137